CLINICAL TRIAL: NCT04506866
Title: Evaluation of InterStim Micro System Performance and Safety (ELITE) to Confirm Long-Term Outcomes - Post Market Clinical Follow-Up Study
Brief Title: InterStim Micro Post Market Clinical Follow-up Study (ELITE)
Acronym: ELITE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the extension of the clinical study duration and to avoid further delaying the reporting of results.
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDT19006
Record Dates: First submitted 2020-08-03; First posted 2020-08-10 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Overactive Bladder; Fecal Incontinence; Non-obstructive Urinary Retention
MeSH Terms: conditions — Urinary Bladder, Overactive; Fecal Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Overactive Bladder Cohort (Other): Subjects with overactive bladder will be treated with InterStim Micro Therapy and followed-up regarding their overactive bladder symptoms.
  Interventions: Device: InterStim Micro
- Fecal Incontinence Cohort (Other): Subjects with fecal incontinence will be treated with InterStim Micro Therapy and followed-up regarding their fecal incontinence symptoms.
  Interventions: Device: InterStim Micro
- Non-Obstructive Urinary Retention Cohort (Other): Subjects with non-obstructive urinary retention will be treated with InterStim Micro Therapy and followed-up regarding their non-obstructive urinary retention symptoms.
  Interventions: Device: InterStim Micro

INTERVENTIONS:
Device: InterStim Micro — Eligible subjects will receive InterStim Micro therapy. Commercial devices will be used within their intended use as described in each geography's approved instructions for use

SUMMARY:
Post-market clinical follow-up for continued assessment of safety and performance to confirm long-term outcomes of the InterStim Micro System for sacral neuromodulation.

ELIGIBILITY:
Overactive Bladder Cohort

Inclusion Criteria:

1. Have a diagnosis of OAB as demonstrated on a 3-day voiding diary with greater than or equal to 8 urgency frequency episodes per day and/or by having a minimum of 3 episodes of urinary urge incontinence in 72 hours
2. Subjects 18 years of age or older
3. Candidate for sacral neuromodulation therapy in accordance with the InterStim Micro System labeling
4. Willing and able to accurately complete study diaries, questionnaires, attend visits, device recharging and comply with the study protocol
5. Willing and able to provide signed and dated informed consent

Exclusion Criteria:

1. Have neurological conditions such as multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury (e.g., paraplegia)
2. Have primary stress incontinence or mixed incontinence where the stress component overrides the urge component
3. Current urinary tract mechanical obstruction (e.g. benign prostatic enlargement or urethral stricture)
4. Have had treatment of urinary symptoms with botulinum toxin therapy in the past 12 months
5. Have knowledge of planned shortwave diathermy, microwave diathermy, or therapeutic diathermy
6. Women who are pregnant or planning to become pregnant
7. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements.
8. Concurrent participation in another clinical study that may add additional safety risks and/or confound study results.

Fecal Incontinence Cohort

Inclusion Criteria:

1. Have a diagnosis of fecal incontinence as demonstrated by a 7-day bowel diary as greater than or equal to 2 incontinent episodes of more than staining (i.e., either slight, moderate or severe soiling)
2. Subjects 18 years of age or older
3. Candidate for sacral neuromodulation therapy in accordance with the InterStim Micro System labeling
4. Willing and able to accurately complete study diaries, questionnaires, attend visits, device recharging and comply with the study protocol
5. Willing and able to provide signed and dated informed consent

Exclusion Criteria:

1. Have neurological conditions such as multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury (e.g., paraplegia)
2. Uncorrected high grade internal rectal prolapse
3. Have knowledge of planned shortwave diathermy, microwave diathermy, or therapeutic diathermy
4. Women who are pregnant or planning to become pregnant
5. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements.
6. Concurrent participation in another clinical study that may add additional safety risks and/or confound study results.

Non-Obstructive Urinary Retention Cohort

Inclusion Criteria:

1. Have a diagnosis of non-obstructive urinary retention as demonstrated by a 7-day urinary voiding diary with a minimum of 5 clean intermittent self-catheterizations
2. Chronic non-obstructive urinary retention with an elevated post-void residual (PVR) that has persisted for at least six months and is documented on two or more separate occasions.
3. Subjects 18 years of age or older
4. Candidate for sacral neuromodulation therapy in accordance with the InterStim Micro System labeling
5. Willing and able to accurately complete study diaries, questionnaires, attend visits, device recharging and comply with the study protocol
6. Willing and able to provide signed and dated informed consent

Exclusion Criteria:

1. Have neurological conditions such as multiple sclerosis, clinically significant peripheral neuropathy or spinal cord injury (e.g., paraplegia)
2. Current urinary tract mechanical obstruction (e.g. benign prostatic enlargement or urethral stricture)
3. Have knowledge of planned shortwave diathermy, microwave diathermy, or therapeutic diathermy .
4. Women who are pregnant or planning to become pregnant
5. Characteristics indicating a poor understanding of the study or characteristics that indicate the subject may have poor compliance with the study protocol requirements.
6. Concurrent participation in another clinical study that may add additional safety risks and/or confound study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mylène Champs, Study Director — Medtronic
Locations (24):
- United States (17):
  - East Coast Institute for Research, Jacksonville, Florida
  - Florida Urology Partners, Tampa, Florida
  - First Urology, Jeffersonville, Indiana
  - Saint Elizabeth Healthcare, Edgewood, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Louisiana State University Health Sciences Center New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Minnesota Urology (Woodbury), Woodbury, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Colon Surgeons of Charleston, Mt. Pleasant, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Urology Partners of North Texas, Arlington, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - West Virginia University, Morgantown, West Virginia
- University Urology Associates, Toronto, Ontario, Canada
- France (2):
  - CHU de Nantes - Hôtel Dieu, Nantes
  - Centre Hospitalier Universitaire De Rennes, Rennes
- Maastricht Universitair Medisch Centrum (MUMC), Maastricht, Netherlands
- Kantonsspital St.Gallen, Sankt Gallen, Switzerland
- United Kingdom (2):
  - Guy's & St Thomas' NHS Foundation Trust - St Thomas' Hospital, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elterman D, Murphy M, Krlin R, Levine R, Yaklic J, Michaels J, Bleier J, Paquette I, Farmer R, Xavier K, Papi B, Wu M, Siproudhis L. Post-Market Study Evaluating Performance of the Rechargeable InterStim Micro System in Fecal Incontinence Patients. Int Urogynecol J. 2025 Apr;36(4):913-921. doi: 10.1007/s00192-025-06127-9. Epub 2025 Apr 5. PMID 40186665

RESULTS

PARTICIPANT FLOW:
Groups:
- Overactive Bladder Cohort: Subjects with overactive bladder were treated with InterStim Micro Therapy and followed-up regarding their overactive bladder symptoms.
- Fecal Incontinence Cohort: Subjects with fecal incontinence were treated with InterStim Micro Therapy and followed-up regarding their fecal incontinence symptoms.
Period: Overall Study
Arm/Group | Overactive Bladder Cohort | Fecal Incontinence Cohort | Non-Obstructive Urinary Retention Cohort
Started | 68 | 53 | 27
Completed | 67 | 52 | 25
Not Completed | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Overactive Bladder Cohort | Fecal Incontinence Cohort | Non-Obstructive Urinary Retention Cohort | Total
Number analyzed (Participants) | 68 | 53 | 27 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (13.2) | 58 (11) | 43 (17.9) | 57 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 48 | 26 | 135
  Male | 7 | 5 | 1 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Number analyzed is different than overall because Race was not collected for sites in EMEA.
  Participants
    White: number analyzed (Participants) | 60 | 44 | 10 | 114
    White | 54 | 37 | 9 | 100
    Black: number analyzed (Participants) | 60 | 44 | 10 | 114
    Black | 5 | 4 | 0 | 9
    Hispanic: number analyzed (Participants) | 60 | 44 | 10 | 114
    Hispanic | 1 | 2 | 0 | 3
    SPANISH/HISPANIC/LATINA: number analyzed (Participants) | 60 | 44 | 10 | 114
    SPANISH/HISPANIC/LATINA | 0 | 1 | 0 | 1
    Asian: number analyzed (Participants) | 60 | 44 | 10 | 114
    Asian | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 12 | 3 | 19
  Netherlands | 0 | 0 | 1 | 1
  United States | 56 | 32 | 7 | 95
  United Kingdom | 0 | 0 | 10 | 10
  France | 8 | 7 | 6 | 21
  Switzerland | 0 | 2 | 0 | 2
Overactive Bladder Quality of Life (OAB-q) Questionnaire Health Related Quality of Life (HRQL) [Mean (Standard Deviation); unit: Total Score] — The Overactive Bladder Quality of Life Questionnaire (OAB-q) is a 33-item validated questionnaire that was developed to assess symptom bother and the impact of overactive bladder (OAB) on health-related quality of life (HRQL). Specifically, The OAB-q consists of an 8-item symptom bother scale and 25-item HRQL scale with 4 domains: coping (8 items), concern/worry (7 items), sleep (5 items) and social interaction (5 items). The score for each of OAB-q domain are summed and transformed to a score ranging from zero to 100. A higher score means a better quality of life. Population: Number analyzed differs from overall because this score applies only to subjects enrolled in the OAB cohort and was not collected for subjects in the FI and the NOUR Cohorts.
  Total Score
    number analyzed (Participants) | 68 | 0 | 0 | 68
    (all) | 44 (21.7) |  |  | 44 (21.7)
Cleveland Clinic Incontinence Score (CCIS) [Mean (Standard Deviation); unit: Score] — Population: Number analyzed differs from overall because this score applies only to subjects enrolled in the FI cohort and was not collected for subjects in the OAB and the NOUR Cohorts.
  Score
    number analyzed (Participants) | 0 | 53 | 0 | 53
    (all) |  | 14 (2.9) |  | 14 (2.9)
Clean intermittent self-catheterizations (CISC) per day [Mean (Standard Deviation); unit: Clean intermittent self-catheterizations] — Population: Number analyzed differs from overall because this measure applies only to subjects enrolled in the NOUR cohort and was not collected for subjects in the OAB and the FI Cohorts.
  Clean intermittent self-catheterizations
    number analyzed (Participants) | 0 | 0 | 27 | 27
    (all) |  |  | 5 (2.3) | 5 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline for HRQL Total Score
Description: The Overactive Bladder Quality of Life Questionnaire (OAB-q) is a 33-item validated questionnaire that was developed to assess symptom bother and the impact of overactive bladder (OAB) on health-related quality of life (HRQL).8 Specifically, The OAB-q consists of an 8-item symptom bother scale and 25-item HRQL scale with 4 domains: coping (8 items), concern/worry (7 items), sleep (5 items) and social interaction (5 items). The score for each of OAB-q domain are summed and transformed to a score ranging from zero to 100.
  We are reporting the change from baseline for HRQL total score. If the change is positive, it means a better quality of life. The higher the positive change is, the better the quality of life is.
Time Frame: 3 months
Population: This score is applicable only for the OAB cohort.
Measure: Mean (Standard Deviation); unit: Total score on a scale
Arm/Group | Overactive Bladder Cohort | Fecal Incontinence Cohort | Non-Obstructive Urinary Retention Cohort
Number analyzed (Participants) | 67 | 0 | 0
Total score on a scale | 33 (24.2) |  |

2. Primary Outcome: Change From Baseline in CCIS Score
Description: The Cleveland Clinic Incontinence Score (Wexner Score) is an established 5-item questionnaire that was developed to assess the frequency and severity of fecal incontinence. CCIS-Wexner score ranges between 0 and 20. Higher scores indicate worse incontinence.
  We are reporting the change from baseline for CCIS Score. If the change is negative, the quality of life improved from baseline. The more negative the score is, the better the quality of life is.
Time Frame: 3 months
Population: This score is only applicable for FI subjects.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Overactive Bladder Cohort | Fecal Incontinence Cohort | Non-Obstructive Urinary Retention Cohort
Number analyzed (Participants) | 0 | 52 | 0
score on a scale |  | -4.06 (3.696) |

3. Primary Outcome: Change From Baseline in the Number of CISC/Day
Description: Subjects reported the clean intermittent self-catheterizations on voiding diaries for 7 consecutive days. We are reporting the change from baseline. If the change is negative, the quality of life is improved from baseline.
Time Frame: 3 months
Population: This measure applies only to subjects in the NOUR Cohort.
Measure: Mean (Standard Deviation); unit: Number of CISC/Day
Arm/Group | Overactive Bladder Cohort | Fecal Incontinence Cohort | Non-Obstructive Urinary Retention Cohort
Number analyzed (Participants) | 0 | 0 | 23
Number of CISC/Day |  |  | -3.52 (2.901)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from consent. We are reporting here the adverse events that started between enrollment (=neurostimulator implant) and exit.
Description: Any adverse event meeting the definition of: serious adverse events and/or adverse device effects were considered reportable for this study.
Arm/Group | Overactive Bladder Cohort | Fecal Incontinence Cohort | Non-Obstructive Urinary Retention Cohort
All-Cause Mortality (participants affected / at risk) | 1/68 | 0/53 | 0/27
Serious Adverse Events (participants affected / at risk) | 3/68 | 8/53 | 4/27
Other Adverse Events (participants affected / at risk) | 5/68 | 8/53 | 14/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overactive Bladder Cohort (N=68) | Fecal Incontinence Cohort (N=53) | Non-Obstructive Urinary Retention Cohort (N=27)
Implant site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Superinfection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overactive Bladder Cohort (N=68) | Fecal Incontinence Cohort (N=53) | Non-Obstructive Urinary Retention Cohort (N=27)
Medical device site discomfort (General disorders) | 1 (1) | 2 (2) | 2 (2)
Implant site pain (General disorders) | 2 (2) | 1 (1) | 4 (4)
Medical device site pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
Device stimulation issue (Product Issues) | 1 (1) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was closed earlier than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT04506866/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT04506866/SAP_001.pdf